CLINICAL TRIAL: NCT02429115
Title: Improving Patient Quality of Life and Caregiver Burden by a Peer-Led Mentoring Program for Patients With Chronic Kidney Disease and Their Caregivers
Brief Title: Peer-mentoring, Quality of Life and Caregiver Burden in Patients With Chronic Kidney Disease and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Nasrollah Ghahramani, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR-1310-07055
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Chronic Kidney Disease
Keywords: peer mentoring; chronic kidney disease; quality of life; pcori; caregiver burden
MeSH Terms: conditions — Renal Insufficiency, Chronic; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Face-to-face peer mentoring (Experimental): Will receive 6 months of face-to-face peer mentoring by a trained peer mentor.
  Interventions: Other: Mentoring
- Online peer mentoring (Experimental): Will receive 6 months of face-to-face peer mentoring by a trained peer mentor.
  Interventions: Other: Mentoring
- Control (No Intervention): Will not receive peer mentoring.

INTERVENTIONS:
Other: Mentoring — Six months of peer-mentoring.
  Arms: Face-to-face peer mentoring; Online peer mentoring

SUMMARY:
Receiving supportive mentoring from well-adjusted individuals who share similar experiences has had a positive influence on adjustment with some chronic diseases. In this study, patients with advanced chronic kidney disease and caregivers of such patients will be randomly assigned to one of three groups: (1) face-to-face PFPP-individuals will receive six months of PFPP peer-mentoring, along with an informational text; (2) online PFPP-individuals will receive six months of online peer-mentoring modeled after the PFPP program, along with an informational text; and (3) information-only control group-individuals will receive the text of the material provided to the other two groups. The study team's decision to include an online version is based on suggestions by previous participants who indicated that this would be convenient for individuals for whom distance and geographic location are major considerations of participation.

The investigators expect that both face-to-face and online peer-mentorship programs will result in improved quality of life among patients with advanced kidney disease and decreased feeling of burden among caregivers of these patients. The investigators also expect that mentorship will lead to improved engagement of patients in their own care.

DETAILED DESCRIPTION:
Chronic kidney disease is very common in the United States, and throughout the world. An increasing number of individuals are diagnosed with late stages of chronic kidney disease, which require treatment with either dialysis or kidney transplant. The number of individuals currently requiring such treatment in the United States is greater than 600,000. Patients with advanced kidney disease and their family members face many challenges in dealing with the disease and the decisions that relate to choice of treatment. Quite frequently, patients and their family members are faced with the need to decide on a treatment option without full awareness of all the options. In such cases, they might make choices with which they will not be satisfied. Poor satisfaction with treatment choice is likely to result in poor quality of life for the patients and increased sense of burden for the caregiver.

Receiving supportive mentoring from well-adjusted individuals who share similar experiences has had a positive influence on adjustment with some chronic diseases. Since 2004, the Kidney Foundation of Central Pennsylvania has conducted a program to formally train patients with kidney disease and their caregivers to become mentors for patients or caregivers who feel they might benefit from such mentoring. The program, the Patient and Family Partner Program (PFPP), was envisioned and designed by a patient with chronic kidney disease and has trained approximately 130 mentors.

In this study, patients with advanced chronic kidney disease and caregivers of such patients will be randomly assigned to one of three groups: (1) face-to-face PFPP-individuals will receive six months of PFPP peer-mentoring, along with an informational text; (2) online PFPP-individuals will receive six months of online peer-mentoring modeled after the PFPP program, along with an informational text; and (3) information-only control group-individuals will receive the text of the material provided to the other two groups. The study team's decision to include an online version is based on suggestions by previous participants who indicated that this would be convenient for individuals for whom distance and geographic location are major considerations of participation.

The investigators expect that both face-to-face and online peer-mentorship programs will result in improved quality of life among patients with advanced kidney disease and decreased feeling of burden among caregivers of these patients. The investigators also expect that mentorship will lead to improved engagement of patients in their own care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage 4 or 5 CKD by a physician / or caregiver to a patient with stage 4 or 5 CKD;
* at least 18 years of age;
* able to read and write in English at the 8th grade level;
* access to computer with internet and email capability

Exclusion Criteria:

* inability to provide consent;
* younger than 18 years of age;
* prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasrollah Ghahramani, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Kidney Foundation of Central Pennsylvania, Harrisburg, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Face-to-face Peer Mentoring Patients; Face-to-face Peer Mentoring Caregivers: Will receive 6 months of face-to-face peer mentoring by a trained peer mentor.
  Mentoring: Six months of peer-mentoring.
- Online Peer Mentoring Patients; Online Peer Mentoring Caregivers: Will receive 6 months of online peer mentoring by a trained peer mentor.
  Mentoring: Six months of peer-mentoring.
- Control Patients; Control Caregivers: Will not receive peer mentoring.
Period: Overall Study
Arm/Group | Face-to-face Peer Mentoring Patients | Online Peer Mentoring Patients | Control Patients | Face-to-face Peer Mentoring Caregivers | Online Peer Mentoring Caregivers | Control Caregivers
Started (Includes patient participants and caregiver participants) | 52 | 52 | 51 | 29 | 29 | 28
Completed | 40 | 42 | 35 | 21 | 22 | 27
Not Completed | 12 | 10 | 16 | 8 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Face-to-face Peer Mentoring Patients | Online Peer Mentoring Patients | Control Patients | Face-to-face Peer Mentoring Caregivers | Online Peer Mentoring Caregivers | Control Caregivers | Total
Number analyzed (Participants) | 52 | 52 | 51 | 29 | 29 | 28 | 241
Age, Customized [Count of Participants; unit: Participants]
  Age ≤ 47 | 11 | 18 | 15 | 7 | 11 | 8 | 70
  47< Age ≤ 54 | 14 | 10 | 12 | 7 | 5 | 6 | 54
  54 <Age ≤ 62 | 12 | 15 | 12 | 9 | 6 | 5 | 59
  62 < Age | 15 | 9 | 12 | 6 | 7 | 9 | 58
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 27 | 31 | 30 | 11 | 9 | 11 | 119
  Female | 25 | 21 | 21 | 18 | 20 | 17 | 122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 26 | 24 | 13 | 13 | 14 | 114
  Non-white | 28 | 26 | 27 | 16 | 16 | 14 | 127
Ethnicity [Count of Participants; unit: Participants]
  Hispanic | 5 | 5 | 7 | 2 | 4 | 2 | 25
  Non-Hispanic | 47 | 47 | 44 | 27 | 25 | 26 | 216
Marital Status [Count of Participants; unit: Participants]
  Married | 16 | 21 | 21 | 20 | 20 | 18 | 116
  Not married | 36 | 31 | 30 | 9 | 9 | 10 | 125
At least some college [Count of Participants; unit: Participants]
  Yes | 22 | 30 | 25 | 11 | 12 | 9 | 109
  No | 30 | 22 | 26 | 18 | 17 | 19 | 132
Employed [Count of Participants; unit: Participants]
  Employed | 13 | 17 | 16 | 11 | 13 | 12 | 82
  Not Employed | 39 | 35 | 35 | 18 | 16 | 16 | 159
Rural [Count of Participants; unit: Participants]
  Rural | 4 | 7 | 9 | 6 | 11 | 8 | 45
  Urban | 48 | 45 | 42 | 23 | 18 | 20 | 196

OUTCOME MEASURES:

1. Primary Outcome: Slope of Change in Kidney Disease Quality of Life-36 Score
Description: The Kidney Disease Quality of Life-36 (KDQOL-36) score is the primary outcome measure. The KDQOL-36 contains 5 subscales: the Physical Component Summary (PCS), Mental Component Summary (MCS), Burden of Kidney Disease (BKD), Symptoms and Problems of Kidney Disease (SPKD), and Effects of Kidney Disease (EKD). The range for the sore of each domain is 0-100. Higher scores represent improved Quality of Life. Change in the scores of components of the KDQOL is the outcome variable of interest. We computed the slopes (rates of change in KDQOL subscales from baseline to 12 months and 18 months) using a random effects ANOVA (random intercept and random slope), and determined if the slopes were different using t-test.
Time Frame: Measured at baseline, at 12 months and at 18 months, slope of change at 18 months reported.
Population: Patient participants.
Measure: Number (95% Confidence Interval); unit: Scores on a scale / Months
Arm/Group | Face-to-face Peer Mentoring Patients | Online Peer Mentoring Patients | Control Patients
Number analyzed (Participants) | 52 | 52 | 51
Scores on a scale / Months
  Effects of Kidney Disease | 2.21 [-1.10 to 5.52] | 4.13 [0.87 to 7.40] | -0.50 [-3.97 to 2.97]
  Burden of Kidney Disease | 3.00 [-1.27 to 7.27] | 5.44 [1.24 to 9.63] | -0.99 [-5.50 to 3.53]
  Short Form-12 Physical Composite | 0.64 [-0.94 to 2.22] | 2.50 [0.95 to 4.06] | -0.70 [-2.36 to 0.97]
  Short Form-12 Mental Composite Score | 1.43 [-0.28 to 3.13] | 3.46 [1.78 to 5.13] | 1.13 [-0.66 to 2.92]
  Symptoms/Problems of Kidney Disease | 3.41 [-0.46 to 6.36] | 6.00 [3.09 to 8.91] | -2.71 [-6.20 to 0.78]
Statistical Analysis 1: Comparison: Face-to-face Peer Mentoring Patients vs Online Peer Mentoring Patients vs Control Patients; Test type: Superiority; p < 0.05, ANOVA

2. Primary Outcome: Slope of Change in Zarit Caregiver Burden Interview (ZBI) Score
Description: The Zarit caregiver Burden Interview (ZBI) score is the primary outcome measure. The score ranges between 0 and 88. Higher scores represent increased caregiver burden (worse outcome); smaller numbers indicate less caregiver burden (better outcome).
  Change in the ZBI score is the outcome variable of interest. We computed the slopes (rates of change in ZBI from baseline to 12 months and 18 months) using a random effects ANOVA (random intercept and random slope), and determined if the slopes were different using t-test.
Time Frame: Measured at baseline, at 12 months and at 18 months, slope of change at 18 months reported.
Population: Caregivers of patients with CKD
Measure: Number (95% Confidence Interval); unit: Scores on a scale / Months
Arm/Group | Face-to-face Peer Mentoring | Online Peer Mentoring | Control
Number analyzed (Participants) | 29 | 29 | 28
Scores on a scale / Months | -2.49 [-5.85 to 0.87] | -3.44 [-6.31 to -0.57] | -1.26 [-4.06 to 1.54]
Statistical Analysis 1: Comparison: Face-to-face Peer Mentoring vs Online Peer Mentoring vs Control; Test type: Superiority; p < 0.05, ANOVA

3. Secondary Outcome: Slope of Change in Patient Activation Measure (PAM)
Description: The Patient Activation Measure (PAM) is the secondary outcome measure. The score ranges between 0-100. Higher scores represent improved patient activation and lower numbers indicate less patient activation. Change in the PAM is the outcome variable of interest. We computed the slopes ( rate of change in the PAM score from baseline to 12 months and 18 months) using a random effects ANOVA (random intercept and random slope), and determined if the slopes were different among the study groups using t-test.
Time Frame: Measured at baseline, at 12 months and at 18 months, slope of change at 18 months reported.
Population: Patient participants
Measure: Number (95% Confidence Interval); unit: Scores on a scale / Months
Arm/Group | Face-to-face Peer Mentoring | Online Peer Mentoring | Control
Number analyzed (Participants) | 52 | 52 | 51
Scores on a scale / Months | 0.95 [-1.96 to 3.86] | 5.66 [2.79 to 8.52] | 0.02 [-3.03 to 3.08]
Statistical Analysis 1: Comparison: Face-to-face Peer Mentoring vs Online Peer Mentoring vs Control; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Face-to-face Peer Mentoring Patients | Online Peer Mentoring Patients | Control Patients | Face-to-face Peer Mentoring Caregivers | Online Peer Mentoring Caregivers | Control Caregivers
All-Cause Mortality (participants affected / at risk) | 3/52 | 4/52 | 5/51 | 1/29 | 1/29 | 1/28
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/51 | 0/29 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/51 | 0/29 | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT02429115/Prot_SAP_000.pdf